CLINICAL TRIAL: NCT03477409
Title: Exposure of NICU Patients to PVC Plasticizers in At-risk Clinical Situation: Biomonitoring Study From Urinary Samples
Acronym: ARMED NEO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-382; 2017-A02073-50 (Other: 2017-A02073-50)
Record Dates: First submitted 2018-02-27; First posted 2018-03-26 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Neonates or Premature Babies; Patient With Urinary Catheter; Patient Hospitalized in NICU
Keywords: plasticizers; medical devices; neonates; exposition
MeSH Terms: conditions — Premature Birth | interventions — Plasticizers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonatal intensive care patients: The purpose of this biomonitoring study consists to evaluate the exposure of newborns and premature babies hospitalized in NICU to these plasticizers (DEHT and TOTM), by qualitative and quantitative measurement of their urinary metabolites
  Interventions: Other: plasticizers

INTERVENTIONS:
Other: plasticizers — The purpose of this biomonitoring study consists to evaluate the exposure of newborns and premature babies hospitalized in NICU to these plasticizers (DEHT and TOTM), by qualitative and quantitative measurement of their urinary metabolites

SUMMARY:
In response to restrictions related to the use of DEHP as a plasticizer for PVC medical devices (MDs), manufacturers have resorted to alternative plasticizers. These are now integrated into many MDs such as infusion sets, extension lines, extracorporeal circuits, nutrition tubings ... etc. The ARMED project (2012-2015) funded by the ANSM, whose goal was to prioritizing the risk linked to the migration of these plasticizers from MDs, has shown that TOTM and DEHT present the best benefit / risk ratio due to lower migration and cytotoxicity. Nevertheless, it is important to evaluate the level of exposure of neonatal intensive care patients, due to the multi exposure to MD made of PVC, the frequent use of intravenous route and the vulnerability of this at-risk population to the metabolites of these plasticizers.

DETAILED DESCRIPTION:
The purpose of this biomonitoring study consists to evaluate the exposure of newborns and premature babies hospitalized in NICU to these plasticizers (DEHT and TOTM), by qualitative and quantitative measurement of their urinary metabolites

ELIGIBILITY:
Inclusion Criteria:

* hospitalized minor patient in NICU
* hospitalized patient in one of the planned services of the study- hospital stay provided for inclusion ≥ 48 hours
* patient with a urinary catheter at the time of inclusion in the study
* patient undergoing during the stay at least 1 of the following medical procedures: enteral nutrition, parenteral nutrition, extra-renal purification, ECMO, transfusion, lipid infusion, plasmapheresis
* patient whose parents have expressed their non-opposition to his participation in the study

Exclusion Criteria:

* death of the patient
* leaving hospital
* patient becoming anuric (diuresis <1mL / kg / h for more than 24 hours) under study

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: minor patient in NICU
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Measurement of urinary levels of DEHT metabolites | at day 1
  The studied metabolites are specific biological markers
Measurement of urinary levels of TOTM metabolites | at day 1
  The studied metabolites are specific biological markers

SECONDARY OUTCOMES:
Correlation of urinary levels of TOTM and DEHT metabolites to corresponding plasticizers doses released by PVC medical devices to which patients are exposed | 18 months after the beginning of the study
  Quantities of plasticizers (TOTM and DEHT) are measured within each MD to which neonates are exposed in NICU. The release doses of plasticizers are evaluated with mathematical model (built from ex vivo experimentations). The study evaluates whether there is a correlation between the doses of TOTM and the DEHT released by the MD and the metabolites levels found in the urine of exposed patients
Comparison of urinary levels of TOTM and DEHT and their metabolites to in vitro cytotoxicity and endocrine disruption and to toxicological data from the literature. | 18 months after the beginning of the study
  The Armed Neo project include laboratory studies to evaluate the cytotoxicity and endocrine disrupting effects of plasticizers and their metabolites. These studies show the concentrations above which DHT, TOTM and metabolites are toxic. The concentrations obtained in the urines of newborns will be compared to these toxicity threshold values

CONTACTS AND LOCATIONS:
Overall Officials: Valérie SAUTOU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France